CLINICAL TRIAL: NCT00699504
Title: A Double Blind, Placebo Controlled, Positive Controlled, Randomized, Crossover Study to Assess the Effect of Cangrelor at the Therapeutic Dose and a Supratherapeutic Dose Level on the QT/QTc Interval in Healthy Volunteers
Brief Title: Assess the Effect of Cangrelor at the Therapeutic Dose and a Supratherapeutic Dose Level on the QT/QTc Interval in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: TMC CAN 08 01
Record Dates: First submitted 2008-06-13; First posted 2008-06-18 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Healthy
Keywords: ECG; QT; Effect of study drug on healthy volunteers
MeSH Terms: interventions — cangrelor; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Lead in Phase (Experimental): Supratherapeutic dose of cangrelor
  Interventions: Drug: cangrelor
- A (Experimental): therapeutic dose cangrelor treatment
  Interventions: Drug: cangrelor
- B (Experimental): supratherapeutic dose cangrelor treatment
  Interventions: Drug: cangrelor
- C (Active Comparator): active comparator treatment
  Interventions: Drug: moxifloxacin
- D (Placebo Comparator): placebo treatment
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: cangrelor — IV bolus 60 mcg/kg; 8 mcg/kg x 3 hrs
  Arms: Lead in Phase
Drug: cangrelor — 30 mcg/kg bolus; 4 mcg/kg/min x 3 hrs. Oral placebo capsule
  Arms: A
Drug: cangrelor — 60 mcg/kg bolus; 8 mcg/kg/min x 3 hrs. Oral placebo capsule
  Arms: B
Drug: moxifloxacin — 400 mg orally. Placebo IV bolus and infusion.
  Arms: C
Drug: placebo — placebo IV and oral
  Arms: D

SUMMARY:
To assess the safety of cangrelor on cardiac repolarization as measured by electrocardiogram (ECG) at therapeutic and supratherapeutic doses.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non pregnant female between 18 years and 45 years of age, inclusive.
2. Female subjects of childbearing potential (ie, who have not undergone a hysterectomy, have not had a tubal ligation, have not been postmenopausal for at least 12 consecutive months, or whose partner has not undergone a vasectomy) must commit either to abstain continuously from heterosexual sexual contact or to use two methods of birth control, one of which must be a barrier method (eg, hormonal contraception, latex condom, diaphragm, or cervical cap), beginning at screening and throughout study participation.
3. A body mass index (BMI) of 19 kg/m2 to 28 kg/m2, inclusive.
4. Agrees to abstain from alcohol consumption for at least 3 days before first dosing with study drug and throughout study participation.
5. Agrees to abstain from caffeine and nicotine replacement therapy during the days of study drug administration and serial ECG measurements.
6. No clinically significant abnormal findings on the physical examination, ECG, blood pressure, heart rate, medical history, or clinical laboratory tests during screening.
7. Serum magnesium and potassium levels within the normal range per the local lab at the time of screening.
8. Healthy volunteer as determined by the screening assessments.
9. Willing and able to comply with all trial requirements.
10. Provide written informed consent before initiation of any study related procedures.

Exclusion Criteria:

1. Known or suspected pregnancy.
2. Increased bleeding risk: ischemic stroke within the last year or any previous hemorrhagic stroke, tumor, or intracranial aneurysm; recent (<1 month) trauma or major surgery; active bleeding.
3. Impaired hemostasis: known International Normalized Ratio (INR) >1.5; past or present bleeding disorder (including congenital bleeding disorders such as von Willebrand's disease or hemophilia, acquired bleeding disorders, and unexplained clinically significant bleeding disorders), thrombocytopenia (platelet count <100,000/µL).
4. Sustained supine systolic blood pressure >140 mmHg or <100 mmHg or a diastolic blood pressure >95 mmHg or <60 mmHg at screening or baseline. Blood pressure may be retested twice in the supine position at intervals of 5 minutes. Blood pressure is considered sustained if either the systolic or the diastolic pressure exceeds the stated limits after three assessments.
5. Resting pulse rate of <50 beats per minute (bpm) or >100 bpm.
6. Abnormality in the 12 lead ECG that, in the opinion of the investigator, increases the risk of participating in the study, such as a corrected QT interval (QTcB or QTcF) >450 milliseconds. The following conduction abnormalities may confound QTc analysis and should be avoided: PR >220 milliseconds, second or third degree atrioventricular (AV) block, intraventricular conduction defect (IVCD) with QRS >120 milliseconds, complete left bundle branch block (LBBB), left anterior fascicular block (LAFB), left posterior fascicular block (LPFB), right bundle branch block (RBBB), or Wolff Parkinson White syndrome (WPW) (WPW defined as PR >120 milliseconds, P axis from 1 to 90, QRS complex >120 milliseconds, delta wave present).
7. Personal history of long QT syndrome, heart failure, or hypokalemia.
8. Personal history of unexplained syncope.
9. Immediate-family history of long QT syndrome.
10. Family history of sudden death.
11. Concurrent medical conditions, therapy, or medications that affect the ECG, especially prolongation of the QT/QTc interval.
12. Use of prescription or over the counter (such as pseudoephedrine containing cold medicines) medication, including herbal remedies and health supplements, known to prolong the QT/QTc interval within 14 days prior to start of the study and throughout study participation.
13. Intention to use prescription (other than thyroid hormone replacement if the dose and regimen of such replacement therapy has been stable for at least 4 weeks prior to screening and is expected to remain stable during study participation or hormonal contraception) or over the counter medication, including herbal remedies and health supplements, within 14 days before the initial dose of study drug and throughout study participation. If this situation arises, inclusion of an otherwise suitable volunteer may be at the discretion of the investigator in discussion with the Sponsor.
14. Current smokers or subjects who have discontinued smoking fewer than 6 months prior to study entry.
15. Donation of any blood or plasma in the last month, or donation of >400 mL of blood within the 3 months preceding study drug administration.
16. Clinically significant abnormalities in clinical laboratory test results.
17. Positive virology screen for human immunodeficiency virus (HIV), hepatitis B, or hepatitis C.
18. Positive urine test for drugs of abuse or alcohol.
19. Clinically significant disease or condition affecting a major organ system, including, but not limited to, gastrointestinal, renal, hepatic, bronchopulmonary, neurological, metabolic or cardiovascular disease.
20. Allergy, hypersensitivity, or contraindication to quinolone antibiotics, cangrelor, or any of their excipients.
21. History of multiple adverse drug allergies of any origin.
22. Deemed by the investigator, for any reason, to be inappropriate for this study, including subjects who are unable to communicate or to cooperate with the investigator.
23. Treatment with other investigational agents or devices within the 30 days preceding randomization, planned use of other investigational drugs or devices during study participation, or previous enrollment in this trial.
24. Inability to give informed consent or high likelihood of being unable to complete the necessary confinement.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2008-06; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in placebo adjusted QTc with the individual correction method (QTcI) following cangrelor administration. | Baseline to treatment

SECONDARY OUTCOMES:
Plasma concentrations of study drug and metabolite | Baseline to treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Charles River Clinical Services NW, Tacoma, Washington, United States

REFERENCES:
- [Derived] Green CL, Whellan DJ, Lambe L, Bellibas SE, Wijngaard P, Prats J, Krucoff MW. Electrocardiographic safety of cangrelor, a new intravenous antiplatelet agent: a randomized, double-blind, placebo- and moxifloxacin-controlled thorough QT study. J Cardiovasc Pharmacol. 2013 Nov;62(5):466-78. doi: 10.1097/FJC.0b013e3182a2630d. PMID 23921301